CLINICAL TRIAL: NCT05868343
Title: Pragmatic Randomized Controlled Trial to Promote Physical Activity Through Home Exercise After Cardiac Rehabilitation
Brief Title: Effectiveness of a Hybrid Cardiac Rehabilitation Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Pamela Tanguay, Principal Investigator, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 101745
Record Dates: First submitted 2023-04-04; First posted 2023-05-22 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiac Rehabilitation; Hybrid; Randomized controlled trial; Physical Activity; Long term
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: First, the centers are randomized to begin the trial period by offering all their patients either hybrid CR or traditional CR. After recruiting half of the target patient population to be included in the study, centers will switch to offering the other type of CR to their new patients admitted from that point on.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Center-based cardiac rehabilitation program (Active Comparator)
  Interventions: Other: Center-based Cardiac Rehabilitation Intervention
- Hybrid cardiac rehabilitation program (Experimental)
  Interventions: Other: Hybrid Cardiac Rehabilitation Intervention

INTERVENTIONS:
Other: Center-based Cardiac Rehabilitation Intervention — The center-based cardiac rehabilitation program is 12 weeks in length. Participants will travel to the center twice a week for the duration of the program. Participants receive an individualized exercise program to be completed at the center according to Canadian recommendations. Twelve pre-recorded educational vignettes on various health topics and two group educational sessions on nutrition are offered to participants in person during the first twelve sessions at the center. In addition, at the beginning of the CR program, participants watch a motivational vignette from one of our patient partners about the importance and benefits of following the CR program. Depending on the needs of each participant, they may be referred to various external clinics within the Vitalité network, such as the Nutrition Service.
  Arms: Center-based cardiac rehabilitation program
Other: Hybrid Cardiac Rehabilitation Intervention — The center-based cardiac rehabilitation program is 12 weeks in length. For the first six weeks, participants are required to attend the hospital twice a week. After that, there will be a gradual increase in home sessions for the remaining six weeks. When a patient has a home session, health professionals follow up with a phone call.Twelve pre-recorded educational vignettes on various health topics and two group educational sessions on nutrition are offered to participants in person during the first twelve sessions at the center. In addition, at the beginning of the CR program, participants watch a motivational vignette from one of our patient partners about the importance and benefits of following the CR program. Depending on the needs of each participant, they may be referred to various external clinics within the Vitalité network, such as the Nutrition Service.
  Arms: Hybrid cardiac rehabilitation program

SUMMARY:
The goal of this pragmatic randomized clinical trial is to compare the effectiveness of a hybrid model of cardiac rehabilitation with a centre-based program in people with cardiovascular disease. The main question it aims to answer is:

• How effective is a hybrid model of CR for people with cardiovascular disease living in a francophone minority community compared to a centre-based model of CR in terms of leading to maintenance of gains (physical activity level, functional capacity, mental health, quality of life) six months after CR? Participants will undergo a 12-week hybrid cardiac rehabilitation program. For the first six weeks, patients will be required to attend the hospital twice a week. After that, there will be a gradual increase in home sessions for the remaining six weeks. When a patient has a home session, health professionals will follow up with a weekly phone call.

Researchers will compare the centre-based cardiac rehabilitation program with the hybrid program to see if the hybrid program can better maintain the level of physical activity, mental health, functional capacity, and quality of life six months after the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Be and adult (over 19 years old)
* Be eligible for Vitalité Health Network Cardiac rehabilitation program.

Exclusion Criteria:

* Have a physical or cognitive condition that precludes participation in an exercise program.
* Have previously participated in a CR program.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 278 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in level of Physical Activity | Questionnaire will be completed at 0 months, 3 months and 9 months
  Description: The Level of Physical Activity will be collected using the International Physical Activity Questionnaire (IPAQ).

SECONDARY OUTCOMES:
Change in health-Related Quality of Life | Questionnaire will be completed at 0 months, 3 months and 9 months
  The Health-Related Quality of life will be collected using the Euro-QoL 5-dimension Questionnaire (EQ-5D-5L). The EQ-5D-5L can be summarized as an index value varying from -0.148 (worst score) to +0.949 (best score).
Change in functional Capacity | Questionnaire will be completed at 0 months, 3 months and 9 months
  The Functional Capacity will be evaluated using the six-minute walk test (6MWT).
Change in anxiety and Depression | Questionnaire will be completed at 0 months, 3 months and 9 months
  Anxiety and depression will be collected using the Hospital Anxiety and Depression Scale (HADS). The total score ranges from 0 to 21 for each subscale (anxiety and depression). A higher score indicates a greater risk of having an anxiety or depression disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Tanguay, Principal Investigator — Université de Sherbrooke
Locations (9):
- Canada (9):
  - Hôpital régional Chaleur, Bathurst, New Brunswick
  - Centre J.K. Irving, Bouctouche, New Brunswick
  - Hôpital Régional de Campbellton, Campbellton, New Brunswick
  - Hôpital de l'Enfant-Jésus RHSJ, Caraquet, New Brunswick
  - Hôpital régional d'Edmundston, Edmundston, New Brunswick
  - Hôpital général de Grand-Sault, Grand Falls, New Brunswick
  - Coeur en santé, Moncton, New Brunswick
  - Hôtel-Dieu Saint-Joseph de Saint-Quentin, Saint-Quentin, New Brunswick
  - Hôpital de Tracadie, Tracadie, New Brunswick

IPD SHARING:
Plan to Share IPD: No